CLINICAL TRIAL: NCT05823870
Title: A Phase 1 Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic Characteristics After Administration of Fixed-dose Combination of DW6014 and Loose Combination of Each Component in Healthy Adult Volunteers in Fasted Condition
Brief Title: This Study is to Compare and Evaluate the Safety and Pharmacokinetic Characteristics (PK) After Administration of DW6014 and Each Component(Empagliflozin and Metformin) in Healthy Adult Volunteers in Fast Condition.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dong Wha Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DW6014-I-1
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — empagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: Empagliflozin and Metformin Period 2: DW6014
  Interventions: Drug: DW6014
- Sequence B (Experimental): Period 1: DW6014 Period 2: Empagliflozin and Metformin
  Interventions: Drug: DW6014

INTERVENTIONS:
Drug: DW6014 — Drug: DW6014 Single oral administration of DW6014 after an overnight fast
  Drug: Empagliflozin and Metformin Combination oral administration of Empagliflozin and Metformin after an overnight fast
  Other Names: Empagliflozin and Metformin

SUMMARY:
This study is to compare and evaluate the safety and pharmacokinetic characteristics (PK) after administration of DW6014 and each component in healthy adult volunteers in fast condition.

DETAILED DESCRIPTION:
This is a Phase 1, randomized, open-label, Oral, Single-dose, two-way crossover study in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged up to 19 years
* Subjects weighing at least 50.0 kg with a BMI between 18.0 kg/m2 and 30.0 kg/m2
* Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination
* Subjects considered eligible for the study participation in accordance to the results of clinical laboratory tests, vital signs, physical examinations and 12-lead ECG conducted at the time of screening, based on the investigational product (IP) characteristics
* Subjects who has a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period

Exclusion Criteria:

* Subjects with any clinically significant hepatic, renal, nervous, respiratory, endocrine, circulatory, tumor, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases or other medical history
* Subject with galactose intolerance, Lapp lactase deficience, glucose-galactose malabsorption or other genetic problem
* Subject following gastrointestinal diseases or gastrointestinal surgery that may affect the absorption of the IP
* Pregnant subjects with a positive urine HCG(human chorionic gonadotropin) test, or lactating female subjects
* Subject with a medical history of hypersensitivity reactions (anaphylaxis or antibiotics etc.) to containing empagliflozin and metformin components, formulation additives, and other drugs (aspirin, antibiotics, biguanide drugs, etc.) or clinically significant hypersensitivity reactions
* Subjects with clinically significant 12-lead ECG findings at the time of screening
* Subjects with a past history of drug abuse or a positive urine drug test
* Subjects with SBP(systolic blood pressure) ≥ 150 mmHg or ≤ 90 mmHg; DBP(diastolic blood pressure) ≥ 100 mmHg or ≤ 60 mmHg; Pulse Rate ≤ 40 bpm or ≥ 100 bpm at the time of screening
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals within 1 months prior to the first IP administration
* Subjects who have administered any prescription drugs or herbal medicines that may affect the characteristics of clinical investigational drugs within 2 weeks prior to the first administration date, or have administered any over-the-counter (OTC) or vitamin preparations within 10 days
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals within 1 months prior to the first IP administration
* Subjects who have participated and were given any other study drugs in other clinical study within 6 months prior to the first IP administration
* Before the first administration date whole blood donation within 2 months or component blood donation within 1 month or received a blood transfusion within 1 month, or the subject who cannot forbid transfusion from the time of obtaining ICF(informed consent form) until PSV(Post-study visit)
* Subjects who have consistently drunk alcohol within 6 months
* Subjects who have smoked more than 10 cigarettes/day on average
* Subjects who have eaten or cannot refrain from eating grapefruit (grapefruit)-containing food from 48 hours before the first administration until the time of PSV(Post-study visit)
* Subjects who have consumed or cannot refrain from consuming caffeine-containing food during the period from 24 hours prior to administration of each period to the time of the last blood sampling
* Subjects who have done and are unable to refrain from strenuous activity
* Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception
* Subjects otherwise considered ineligible for participation due to other reasons including clinical laboratory test results not mentioned in the inclusion/exclusion criteria at the investigator's discretion

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
AUC0-t | 48 hour
  AUC0-t of Empagliflozin and Metformin
Cmax | 48 hour
  Cmax of Empagliflozin and Metformin

SECONDARY OUTCOMES:
Tmax | 48 hour
  Tmax of Empagliflozin and Metformin
AUCinf administration to infinity) | 48 hour
  AUCinf of Empagliflozin and Metformin
t1/2 | 48 hour
  t1/2 of Empagliflozin and Metformin
CL/F | 48 hour
  CL/F of Empagliflozin and Metformin
Vd/F | 48 hour
  Vd/F of Empagliflozin and Metformin

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea